CLINICAL TRIAL: NCT03040557
Title: Therapeutic Effect of Minimalist Flexible Footwear and Insoles on Clinical, Functional and Biomechanical Aspects of the Individuals With Plantar Fasciitis and Calcaneus Spur
Brief Title: Flexible Footwear and Insole in Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Paula Ribeiro, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APRibeiro
Record Dates: First submitted 2016-10-01; First posted 2017-02-02 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Plantar Fasciitis of Right Foot (Disorder); Heel Spur
Keywords: plantar fasciitis; shoes; insoles; pain; foot
MeSH Terms: conditions — Heel Spur; Fasciitis, Plantar; Pain

STUDY DESIGN:
Intervention Model Description: A randomized, parallel and controlled clinical trial with blind assessor was conducted in which 79 women were randomized and allocated to the intervention groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention groups were: minimalist flexible footwear group-MFG (n=12 women with PF; n=15 women with CS), Orthopedic insole on minimalist footwear group-COIG (n=14 women with PF; n=14 women with CS) and control-GC group (n=24). Both groups were followed for six months and were assessed at baseline condition and after three and six months (end of intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible footwear (Active Comparator): The intervention with flexible footwear in women with plantar fasciitis (MFG), acute n=12 and chronic=15) will have a duration will be six months, for six hours a day, seven days a week (42 hours / week).
  Interventions: Device: Flexible footwear
- Orthopedic insole (Active Comparator): The intervention with orthopedic insole in women with plantar fasciitis (COIG, acute n=14 and chronic=14) will have a duration will be six months, for six hours a day, seven days a week (42 hours / week).
  Interventions: Device: Orthopedic insole

INTERVENTIONS:
Device: Flexible footwear — - Arm Flexible footwear: The intervention will be with flexible shoes in women with plantar fasciitis (acute and chronic) and will have a duration will be six months, for six hours a day, seven days a week (42 hours / week).
  Arms: Flexible footwear
Device: Orthopedic insole — - Arm Orthopedic insole: The intervention will be with orthopedic insole in women with plantar fasciitis (acute and chronic) and will have a duration will be six months, for six hours a day, seven days a week (42 hours / week).
  Arms: Orthopedic insole

SUMMARY:
The plantar fasciitis (PF), most frequent injury of the musculoskeletal system, is the main cause of heel pain and functional disability. The mechanical stress, stretching of plantar fascia consequently the overload on the feet, is a major intrinsic causes the onset of FP, especially when exposed to repetitive activities, such as walking. Another extrinsic etiologic factor of great influence is inadequate shoes that can lead to a deterioration and progression of the disease. One of the great difficulties of their conservative treatment is long rehabilitation period, lasting on average 10 to 18 months. Among them, the insoles stand out as one of the effective mechanical treatments to improve the immediate pain symptoms, in the short term. Other literary evidence, not specific to FP, has shown the benefits, the short and long term, a flexible footwear promotes more flexible feet and overload reduction. Objective: Verify therapeutic effect in the long term, a flexible footwear and low cost and orthopedic insole on the clinical aspect, functional and biomechanics of the gait of women with acute FP and chronic with presence of heel spur. It will be conducted a randomized controlled trial with blinded evaluator, in which 79 women with plantar fasciitis will be randomized and allocated to the intervention group with minimalist flexible footwear (MFG, acute n=12 and chronic=15) or the intervention group with orthopedic insole (COIG, acute n=14 and chronic n=14) or control group (CG, n=24). The intervention will have duration six months, six hours a day, seven days a week (42 hours/week). For all groups will be allowed to use pain medication support (paracetamol 500 mg) with a maximum dose of two grams daily. The primary outcome will be the symptom of pain verified by visual analogue scale (VAS), the inability to areas of the feet by the total score of the FFI (Foot Function Index), health feet by FHSQ-Br questionnaire (Foot Health Questionnaire Status) and the distance traveled by the six-minute walk test (6MWT). The secondary: plantar pressure and ground reaction force during gait, paracetamol consumption and the joint angles of the lower limbs. The effects of time (Start, 3 and 6 months), group (GIC and GIP CG) and interaction (time and group) are calculated by means of ANOVA case-wise two factors. A 5% alpha to significant differences and Cohen coefficient for describing the size effect of the intervention is assumed.

DETAILED DESCRIPTION:
A prospective controlled study with random allocation. The independent variable (group) has three levels: intervention with flexible footwear, intervention with custom orthopedic insoles and control without intervention, only with medical conservative treatment. This independent variable is related to the set of dependent variables stemmed from clinical, functional and biomechanical data. All groups, both will use the intervention minimalist flexible footwear (MFG), as the intervention group insole (COIG) and the group that did not receive intervention (GC) shall consist of patients with PF (plantar fasciitis) in different stages of the disease.These will be required to fit in all the pre-established criteria for diagnosis of the disease confirmed by physical examination, X-ray and ultrasound. Patients in the group with chronic fasciitis plantar associated with heel spur should necessarily present themselves diagnosed radiographically by the doctor that came in the Rheumatology Clinic of the University. All participants will be informed of the procedures in this research through a free and informed consent form, prepared in accordance with Resolution 466/12 of the National Health Board. The eligibility criteria for this study will be: female volunteers aged between 30 and 50 years, body mass index (BMI) less than 35 kg / m2, no history of any surgical procedure on knees, ankles and hips or muscle injury in the last 6 months and no neurological and rheumatologic disease diagnosed. Furthermore, they may not show difference in length of the lower limbs greater than 1 cm and rigid hallux and performing some kind of conservative treatment for PF, except drug. Patients should be able to walk independently for at least 6 hours a day without the aid of orthotics / canes to perform their activities of daily living. There may also have prostheses and / or orthoses in the lower limbs. Patients may not have received corticosteroid injection in the heel in previous periods of three and six months, respectively. In addition to these criteria, patients may not present: joint instability ankle (positive test results of the medial ligament and lateral), dementia or inability to provide information consistent.It will be conducted a randomized controlled trial with blinded evaluator, in which 75 women with plantar fasciitis will be randomized and allocated to the intervention group with flexible footwear (MFG, acute n=15 and chronic=15) or the intervention group with orthopedic insole (COIG, acute n=15 and chronic n=15) or control group (CG, n=15). The intervention will have duration six months, six hours a day, seven days a week (42 hours/week). For all groups will be allowed to use pain medication support (paracetamol 500 mg) with a maximum dose of two grams daily. The primary outcome will be the symptom of pain verified by visual analogue scale (VAS), the inability to areas of the feet by the total score of the FFI (Foot Function Index), health feet by FHSQ-Br questionnaire (Foot Health Questionnaire Status) and the distance traveled by the six-minute walk test (6MWT). The secondary: plantar pressure and ground reaction force during gait, paracetamol consumption and the joint angles of the lower limbs. The effects of time (Start, 3 and 6 months), group (GIC and GIP CG) and interaction (time and group) are calculated by means of ANOVA case-wise two factors. A 5% alpha to significant differences and Cohen coefficient for describing the size effect of the intervention is assumed.

ELIGIBILITY:
Inclusion criteria:

* Women volunteers aged between 30 and 50 years
* Diagnosis of plantar fasciitis (PF) or heel spur
* Healthy women
* Body mass index (BMI) less than 35 kg/m2

Exclusion criteria:

* Difference in length of the lower limbs greater than 1 cm
* Surgical procedure on the knees, ankles and hips or muscle injury in the last 6 months
* Diagnosed neurological and rheumatic disease
* Rigid hallux
* Conservative treatment for PF, except drug
* Walk dependent with prostheses and / or orthoses in the lower limbs
* Corticosteroid injection in the heel in previous periods of three and six months, respectively
* Joint instability ankle
* Dementia or inability to provide information consistent

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Symptom pain on foot | Change from Symptom pain on foot at 3 and 6 months
  The primary outcome will be the symptom of pain verified by visual analogue scale (VAS/cm)
Foot Function Index (FFI) | Change from domains of the FFI at 6 months
  The domains of disability feet by the all score of the FFI (Foot Function Index in score)
Foot Health Status Questionnaire (FHSQ-Br) | Change from FHSQ-Br at 6 months
  Health feet by FHSQ-Br questionnaire (Foot Health Status Questionnaire in units)
Six-minute walk test (6MWT) | Change from 6MWT at 3 and 6 months
  The distance traveled by the six-minute walk test (6MWT in kilometers)

SECONDARY OUTCOMES:
Plantar pressure | Change from plantar pressure at 3 and 6 months
  The peak pressure (kPa), contact area (cm) and contact time (ms) by platform pressure
Ground reaction force | Change from maximum force at 3 and 6 months
  Maximum Force (Newton/N) during gait
For all groups will be allowed to use pain medication support for foot pain | The groups will be allowed to use pain medication support for foot pain at 3 and 6 months
  For all groups will be allowed to use pain medication support (paracetamol 500 mg) with a maximum dose of two grams daily.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula Ribeiro, Ph.D., Principal Investigator — University of the São Paulo
Locations (1):
- School of Medicine, University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ribeiro AP, de Souza BL, Joao SMA. Effectiveness of mechanical treatment with customized insole and minimalist flexible footwear for women with calcaneal spur: randomized controlled trial. BMC Musculoskelet Disord. 2022 Aug 13;23(1):773. doi: 10.1186/s12891-022-05729-4. PMID 35964021